CLINICAL TRIAL: NCT01398423
Title: A 12 Week, Phase II Trial of the Safety, Pharmacokinetics, and Efficacy of INV-144 Compared With Losartan Potassium in Patients With Hypertension and Type 2 Diabetes Mellitus With Nephropathy
Brief Title: INV-144 Versus Losartan in Hypertension and Type 2 Diabetes Mellitus Patients With Macroalbuminuria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: InVasc Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INV144-201
Record Dates: First submitted 2011-07-19; First posted 2011-07-20 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Hypertension; Diabetes Mellitus, Type 2
Keywords: Hypertension; Diabetes mellitis; Nephropathy; Albuminuria
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2; Kidney Diseases; Albuminuria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active control (Active Comparator): Losartan potassium (50 mg) plus placebo to match alpha lipoic acid (600 mg)
  Interventions: Drug: Active Control
- INV-144 (Experimental): INV-144 is a combination drug product consisting of losartan potassium (50mg) and alpha lipoic acid (600 mg)
  Interventions: Drug: INV-144

INTERVENTIONS:
Drug: Active Control — Losartan potassium (50 mg) plus placebo to match alpha lipoic acid (600 mg)
  Arms: Active control
Drug: INV-144 — INV-144 is a combination drug product consisting of losartan potassium (50mg) and alpha lipoic acid (600 mg)
  Arms: INV-144

SUMMARY:
A randomized, double-blind, active control trial to determine the safety, efficacy and pharmacokinetics of INV-144 versus losartan potassium plus placebo in subjects with hypertension and Type 2 diabetes mellitus with nephropathy as evidenced by albuminuria.

DETAILED DESCRIPTION:
A multicenter, randomized, double-blind, parallel-group, active-control trial is designed to evaluate the safety and efficacy of INV-144 versus losartan plus placebo co-administered once daily for 12 weeks in subjects who have type 2 diabetes and hypertension with nephropathy as evidenced by albuminuria.

Approximately 92 adult subjects will be enrolled and randomized in a 1:1 ratio to receive either INV-144 or losartan plus placebo once daily for 12 weeks. The goal is to have approximately 80 subjects complete the entire study.

The trial will consist of a 4-week open-label losartan run-in period, a 12-week double-blind active treatment period, and a 4-week safety follow-up period. Efficacy will be evaluated by measurement of UACR, systolic and diastolic blood pressure, and the HOMA-IR ratio. Safety will be monitored throughout the study by evaluation of adverse events (AEs), physical examinations (PEs), clinical laboratory results, vital signs, and electrocardiograms (ECGs).

Blood samples for PK analysis will be obtained in a subset of approximately 22 subjects, at 2 to 4 sites, to ensure that PK data are obtained from a minimum of 9 subjects in each treatment arm.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women, 18 to 85 years of age, inclusive.
2. Able and willing to understand and provide written informed consent.
3. Documented hypertension defined by 1 of the following:

   Currently treated with antihypertensive medications, or Untreated with a seated systolic blood pressure (mean of 3 readings) between 126 and 180 millimeters of mercury (mm Hg).
4. Documented type 2 diabetes mellitus defined by 1 of the following:

   Currently treated with anti-diabetic medication (oral and/or insulin), or Fasting serum glucose level ≥126 mg/dL.
5. Documented nephropathy evidenced by a UACR of 300 to 3000 mg/g.
6. Both men and women of child bearing potential (i.e., not surgically sterile or post-menopausal defined as age >40 years without menses for ≥2 years) must agree to use 1 of the following forms of reliable contraception:

Abstinence, meaning a total lack of sexual activity, Oral contraceptives ("the pill") or other hormonal contraceptive methods, Intrauterine device, Double-barrier method (diaphragm or condom plus spermicidal cream), or If female, male partner sterilization.

Exclusion Criteria:

1. Required use of an ACE inhibitor, ARB, direct renin inhibitor, or aldosterone antagonist other than study drug, while on the study.
2. Systolic blood pressure >180 mm Hg (mean of 3 seated readings, 5 minutes apart, using the subject's dominant arm).
3. Chronic kidney disease stage 4 or higher defined as an estimated glomerular filtration rate <30 mL/min per 1.73 m2 (abbreviated MDRD equation).
4. Hepatic impairment defined by serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST)>2 x the upper limit of normal.
5. Diagnosis of type 1 diabetes or non-diabetic renal disease, including but not limited to renal-artery stenosis, primary glomerular disease, autoimmune renal diseases, etc.
6. Severe anemia defined as hemoglobin < 8 g/dL.
7. Congestive heart failure with New York Heart Association Class II, III, or IV symptoms.
8. Thiamine (Vitamin B1) deficiency or known alcohol abuse within the past year. If alcohol abuse is suspected, subject must have a normal thiamine blood level documented prior to study entry.
9. Any radiocontrast-facilitated study within 30 days prior to Study Day 1.
10. Cerebrovascular accident within the previous 6 months, or have had a transient ischemic attack within the previous year.
11. Pregnant or nursing women; women of childbearing potential must have a negative serum pregnancy test at Screen.
12. Known adverse reaction to losartan and/or ALA.
13. Participation in another clinical trial or have received an investigational agent for any reason within 30 days of Study Day 1.
14. Any other condition that in the opinion of the Investigator, may adversely affect the safety of the subject, the subject's ability to complete the study, or the outcome of the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2011-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Safety | 12 weeks
  Safety will be monitored throughout the study by evaluation of adverse events (AEs), physical examinations (PEs), clinical laboratory results, vital signs, and electrocardiograms (ECGs).

SECONDARY OUTCOMES:
Efficacy | 12 weeks
  Efficacy will be evaluated by measurement of UACR, systolic and diastolic blood pressure, and the HOMA-IR ratio.

CONTACTS AND LOCATIONS:
Overall Officials: William Schaeffer, Study Director — InVasc Therapeutics, Inc.
Locations (18):
- United States (18):
  - Garden Grove, California
  - La Mesa, California
  - Northridge, California
  - Riverside, California
  - Tustin, California
  - Kissimmee, Florida
  - Miami, Florida
  - Macon, Georgia
  - Tucker, Georgia
  - Reisterstown, Maryland
  - Brooklyn Center, Minnesota
  - Cary, North Carolina
  - Greenville, North Carolina
  - New Bern, North Carolina
  - Raleigh, North Carolina
  - Aiken, South Carolina
  - San Antonio, Texas
  - Norfolk, Virginia